CLINICAL TRIAL: NCT07134231
Title: In Situ Evaluation of the Anti-cavity Efficacy of Three Dentifrices Using an Intra-oral Enamel Demineralization-Remineralization Model
Brief Title: Clinical Study to Evaluate the Anti-cavity Efficacy of Three Dentifrices: An In Situ Model
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Collaborators: Federal University of Alagoas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: CRO-2025-08-DEMI-REMI-BZ-CB
Record Dates: First submitted 2025-08-14; First posted 2025-08-21 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-08

CONDITIONS: Demineralization; Remineralization; Dental Cavity; Enamel Lesions
Keywords: enamel mircrohardness; enamel demineralization-remineralization
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Intervention Model Description: This is a Phase III, randomized, one-center, crossover group, triple blind, clinical study with an intra-oral enamel Demineralization - Remineralization In-Situ Model.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Test Group (Experimental): Subjects will brush using a fluoride free toothpaste in a chalk base with herbal ingredients and a soft bristle toothbrush
  Interventions: Drug: Fluoride free toothpaste in a chalk base; Device: Toothbrush
- Positive Control Group (Active Comparator): Subjects will brush using a fluoride toothpaste containing 1000 ppm MFP and 1.5% arginine in a PCC/RNCC base and a soft bristle toothbrush
  Interventions: Drug: Fluoride Toothpaste; Device: Toothbrush
- Negative Control Group (Sham Comparator): Subjects will brush using a fluoride free toothpaste in a PCC/RNCC base and a soft bristle toothbrush
  Interventions: Drug: Fluoride free toothpaste in a PCC/RNCC base; Device: Toothbrush
- Washout Group (Other): Subjects will brush using a fluoride free toothpaste in a PCC/RNCC base and a soft bristle toothbrush for 9 days, between the treatment phases.
  Interventions: Drug: Fluoride free toothpaste in a PCC/RNCC base; Device: Toothbrush

INTERVENTIONS:
Drug: Fluoride free toothpaste in a chalk base — Fluoride free toothpaste in a chalk base with herbal ingredients
  Arms: Test Group
Drug: Fluoride Toothpaste — Fluoride toothpaste containing 1000 ppm MFP and 1.5% arginine in a PCC/RNCC base
  Arms: Positive Control Group
Drug: Fluoride free toothpaste in a PCC/RNCC base — Fluoride free toothpaste in a PCC/RNCC base
  Arms: Negative Control Group; Washout Group
Device: Toothbrush — A commercially available adult soft bristle toothbrush

SUMMARY:
Clinical study to evaluate the anti-cavity effectiveness of three dentrifices using an intra-oral enamel Demineralization and Remineralization In-Situ Model. This is a six-week duration, Phase III, single-center, triple-blind crossover study. Thirty-six healthy adults will be randomly allocated to three groups for the treatment phases, which are interspersed with washout periods.

DETAILED DESCRIPTION:
This Phase III, randomized, triple-blind, crossover study will assess the anti-cavity effectiveness of three different dentrifices. Thirty-six participants, aged 18-70, will use an intra-oral appliance. For six weeks, they will be divided into three treatment groups and instructed to brush twice daily with one of the following: one using a fluoride-free toothpaste with a chalk base and herbal ingredients, another using a fluoride toothpaste containing 1000 ppm MFP and 1.5% arginine in a PCC/RNCC base, and a negative control group using a fluoride-free toothpaste in a PCC/RNCC base. Each participant will receive a soft-bristle toothbrush and the toothpastes assigned.

Between each five-day treatment phase, participants will have a nine-day washout period, using a fluoride-free toothpaste in a PCC/RNCC base. The study's eight-visit schedule includes a baseline visit, three treatment phases, three washout periods interspersed between the treatment phases, and a final visit. The primary outcome will be the measurement of changes in enamel microhardness, with assessments taking place both before and after each treatment to determine the impact on the enamel. The expected outcome is the confirmation of the alternative hypothesis, which predicts a reduction in the percentage of mineral loss from the surface of bovine enamel after using dentifrices containing 1000 ppm MFP with 1.5% arginine or herbal ingredients for five days each, compared to the control group. The percentage of mineral loss on the tooth surface relative to baseline will be used to quantify the extent of reduction in enamel demineralization. A two factor ANCOVA using the baseline as the covariate will be conducted to determine if a significant treatment effect exists. Adverse events and compliance will be closely monitored, with strict confidentiality maintained for all participants.

ELIGIBILITY:
Inclusion Criteria: Potential subjects must meet ALL of the following criteria:

* Males and females, between 18-70 years of age (inclusive);
* Informed Consent Form signed and availability for the duration of the study;
* Good general health (absence of any condition that, in the opinion of the Principal Investigator, might constitute a risk to the subject while participating in the study. Examples include heart problems, valve/hip replacements, etc);
* Willingness to provide information related to their medical history;
* Minimum of 20 uncrowned permanent natural teeth (excluding third molars); Normal salivary flow;
* Willingness to wear an intra-oral appliance all day as instructed except when eating and drinking.

Exclusion Criteria: Potential subjects must NOT HAVE ANY of the following conditions:

* Oral pathology, chronic disease, or a history of allergy to testing products;
* Subject using anticonvulsants, antihistamines, antidepressants, sedatives, tranquilizers, anti-inflammatory medication or daily analgesics within one month prior to the start of the study or scheduled to start such intake during the course of the study;
* Subject participating in any other clinical study;
* Subject pregnant or breastfeeding;
* Subject allergic to oral care products, personal care consumer products, or their ingredients;
* Extended use of antibiotics or therapeutic mouthwash any time during the three months prior to entry into the study;
* A medical history reporting that the subject has a current systemic or autoimmune disease, such as diabetes, lupus, etc.;
* Ongoing use of medications known to affect the gingival tissues (i.e. calcium channel blockers, phenytoin, cyclosporine);
* Advanced periodontal disease (purulent exudate, tooth mobility, and/or extensive loss of periodontal attachment or alveolar bone). Pocket depth equal or greater than 4 mm;
* Five or more decayed, untreated dental sites (cavities);
* Current smokers and subjects with a history of alcohol or drug abuse;
* Dental work prevents wearing of the appliance or a reported need to wear a night guard.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2025-10-09 (Actual); Primary Completion 2025-12-11 (Actual); Study Completion 2025-12-11 (Actual)

PRIMARY OUTCOMES:
Microhardness change | 6 weeks
  The primary outcome of this study will be the change in the hardness of an intra-oral appliance before and after treatment. It will be determined by measuring the length of an indentation made on the appliance, which in turn allows for the calculation of its hardness value. The effectiveness of the treatment in reducing enamel demineralization by quantifying the percentage of mineral loss relative to the baseline will also be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Natanael Santos, PhD, Principal Investigator — Federal University of Alagoas
Locations (1):
- Federal University of Alagoas, Maceió, Alagoas, Brazil

IPD SHARING:
Plan to Share IPD: No